CLINICAL TRIAL: NCT02637154
Title: The Effect of Motivational Interview and Intensive Education on HbA1C Values and Glucose Variability in Adolescents With Poorly Controlled Type 1 Diabetes
Brief Title: Motivational Interview in Adolescents With Poorly Controlled Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mari Pulkkinen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MoHa
Record Dates: First submitted 2015-12-10; First posted 2015-12-22 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Adolescent; Type 1 diabetes; Metabolic control; Motivational interviewing
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Active Comparator): With 30 patients Motivational Interviewing method will be used during each visit
  Interventions: Behavioral: Motivational Interviewing
- Standard Education (Active Comparator): With 30 patients Standard Education material will be used during each visit
  Interventions: Behavioral: Standard Education

INTERVENTIONS:
Behavioral: Motivational Interviewing — Motivational Interviewing method
  Arms: Motivational Interviewing
Behavioral: Standard Education — Standard Education material will be used
  Arms: Standard Education

SUMMARY:
This study investigates the effect of motivational interviewing and intensive education on HbA1c values and glucose variability in poorly controlled adolescent T1D patients.

In the present study motivational interviewing (MI) will be integrated to clinicians' daily practice, as a part of normal clinical visit. In this randomized, controlled trial hypothesis is, that applying motivational interviewing during regular clinical visits results in better acceptance and subsequently enhanced metabolic control in adolescents with poorly controlled type 1 diabetes.

DETAILED DESCRIPTION:
Background Type 1 diabetes (T1D) patients with optimal glycemic control suffer markedly less from long term diabetic complications than those with poor control. Increased glycohemoglobin (HbA1C) levels predict the complication risk. The development of diabetic complications seems to accelerate during puberty, and poor metabolic control during adolescence or young adulthood markedly increases the incidence of micro- or macrovascular complications during subsequent years. On the other hand, intensive treatment during adolescence has been reported to reduce the risk of microvascular complications, even if the control later on becomes poorer. This implicates that interventions targeting at improved glycemic control during adolescence probably have sustained beneficial effects on the overall morbidity in patients T1D.

The glycemic control of Finnish adolescents with T1D is poor. Insulin resistance and impaired metabolic control are common problems. Treatment of the disease during puberty can be complicated and particularly treatment adherence often declines in youth. Inexpensive and easily adoptable methods for clinicians are needed to overcome treatment problems faced with adolescent patients.

At present, there are no generally recommended approaches for clinicians to apply in order to motivate adolescents with poor glycemic control towards better treatment adherence. To this end, motivational interviewing (MI) has been used to an increasing degree in health care professionals in the treatment of variety of disorders and behavioral problems, such as alcohol and drug problems, gambling, and cardiovascular diseases. Motivational interviewing is a counseling approach designed to facilitate intrinsic motivation in the patient to change behavior. Significant body of evidence supports the view that MI improves commitment to care when added to other treatment. However, only a few studies have evaluated MI in the treatment of adolescent diabetes patients, with outcomes ranging from substantial benefit to neutral. MI is a promising approach for the treatment adolescent type 1 diabetics but there is a clear demand for methodologically solid studies.

Aims The aim of the present study is to investigate the effect of motivational interviewing and intensive education on HbA1c values and glucose variability in poorly controlled adolescent T1D patients. Secondarily, it will be investigated whether improved glycemic control is associated with improvements in vascular parameters, metabolic markers, markers of bone health and health related quality of life.

Hypothesis In the present study motivational interviewing (MI) will be integrated to clinicians' daily practice, as a part of normal clinical visit. In this randomized, controlled trial hypothesis is, that applying motivational interviewing during regular clinical visits results in better acceptance and subsequently enhanced metabolic control in adolescents with poorly controlled type 1 diabetes.

Study protocol All physicians participating in the study are trained to use standardized educational (SE) material. In addition half of the physicians are randomized to motivational interview (MI) group. They are trained by professor Martti Tuomisto's group to use MI in a one day workshop with refresher practical rehearsal course prior to study start. To secure that MI is sufficiently applied, the physician/patient discussions will be monitored by the Tuomisto group. All researchers randomized to the MI group will receive continuous feedback from the Tuomisto group on their performance (i.e. level of applying MI) and if needed re-trained for MI.

Patients with Hba1c > 75 mmol/mol are identified from hospital records, and are considered eligible for the current study. The patients willing to participate are randomized either to MI plus SE or SE group.

Study Protocol Every visit includes a physical examination (including evaluation of the stage of puberty and testis volume at the start and at 12 months), measurement of height, weight, growth velocity, body mass index (BMI), blood pressure and waist circumference, usage of SE material, and in the MI group usage of MI during the patient visit. The intervention in the MI group consists of a MI type of introduction at the beginning of each patient visit, and applying MI principles and procedures on each educational item discussed during the patient visit. Adherence to MI intervention protocols will be checked using recorded samples of therapy interactions. HbA1c levels are also measured in every visit.

Six days blinded continuous glucose monitoring will be performed at baseline and during the follow-up (0, 6 and 12 months).

Fasting venous blood samples are obtained at baseline and at 12 months. Investigators will evaluate health related quality of life (QoL) in study participants at baseline, and at completion of the study.

Dual- energy x-absorptiometry (DXA) is performed at baseline and at 12 months. Vascular assessments will be performed at baseline and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of type 1 diabetes with at least 2 years duration and HbA1c > 75 mmol/mol on two consecutive visits, age 12-15.9 years and pubertal (Tanner) stage 2 or more at inclusion

Exclusion Criteria:

* celiac disease with poor control; diagnosis of psychiatric disease; and other chronic disease requiring per oral glucocorticoid treatment

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C values (mmol/mol) | 12 months
  HbA1c levels (mmol/mol) are measured in every visit (AfinionTM).
Change in glycaemic variability | 12 months
  Six days blinded continuous glucose monitoring (CGM) (iPro, Medtronic) will be performed at baseline and during the follow-up. Blinded CGM curves (0 and 12mo) will be analyzed to study effect on glycemic variability. Standard deviation (SD) of blood glucose values and mean amplitude of glycemic excursions (MAGE) will be used as parameters to define glycemic variability.

SECONDARY OUTCOMES:
Influence of changes in markers of vascular health (IMT) | 12 months
  The association between glycemic control and vascular wall morphology is assessed by imaging of the carotid, femoral, brachial and radial artery intima media thickness (IMT as millimeters - mm:s) with ultrasound. Results will be compared to previously established measurements from healthy children. Vascular assessment will be performed at baseline and at study completion.
Influence of changes in markers of vascular health (PWV) | 12 months
  The association between glycemic control and central and peripheral arterial thickness is assessed with pulse wave velocity (PWV - as meters / second - m/s) using applanation tonometry. Results will be compared to previously established measurements from healthy children. Vascular assessments will be performed at baseline and at study completion.
Influence of changes in bone mineral density (BMD) | 12 months
  Dual- energy x-absorptiometry (DXA) is performed at baseline and at 12 months for analyses of BMD (total body less head, lumbar spine) and body composition, using the Hologic Discovery device (indicated as SD of Z-score).
Influence of changes in quality of life | 12 months
  Health related quality of life (QoL) in study participants will be evaluated at baseline, and at completion of the study with the KINDL-R questionnaires
Influence of changes in markers of inflammation (IL-6 - pg/ml) | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for later analysis of serum inflammatory marker serum IL-6.
Influence of changes in markers of inflammation (high-sensitive-c-reactive-protein CRP - mg/l). | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for later analysis of serum inflammatory marker hs-CRP.
Influence of changes in insulin-like-growth-factor IGF-I levels | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for later analysis of serum insulin-like-growth-factor IGF-I (ng/ml) levels.
Influence of changes in markers of bone turnover (serum aminoterminal propeptide of type I collagen (PINP - ng/ml)). | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for later analysis of markers of bone turnover (PINP - ng/ml).
Influence of changes in vitamin D status (25-hydroxy-D) ng/ml | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for analysis of changes in vitamin D status.
Influence of changes in marker of bone turnover: osteocalcin (ng/ml) | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for analysis of changes in bone turnover marker osteocalcin.
Influence of changes in marker of bone turnover: aminoterminal telopeptide of type I collagen (INTP - ng/ml) | 12 months
  Fasting venous blood samples are obtained at baseline and at 12 months for analysis of changes in bone turnover marker INTP.

CONTACTS AND LOCATIONS:
Overall Officials: Mari Pulkkinen, MD PhD, Principal Investigator — Specialist in Pediatric Endocrinology
Locations (3):
- Finland (3):
  - Helsinki University Central Hospital, Pediatric Diabetes Unit Espoo, Espoo
  - Helsinki University Central Hospital, Pediatric Endocrinology Unit, Helsinki
  - Oulu University Hospital, Pediatric Endocrinology Unit, Oulu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group; Nathan DM, Zinman B, Cleary PA, Backlund JY, Genuth S, Miller R, Orchard TJ. Modern-day clinical course of type 1 diabetes mellitus after 30 years' duration: the diabetes control and complications trial/epidemiology of diabetes interventions and complications and Pittsburgh epidemiology of diabetes complications experience (1983-2005). Arch Intern Med. 2009 Jul 27;169(14):1307-16. doi: 10.1001/archinternmed.2009.193. PMID 19636033
- [Background] Bryden KS, Dunger DB, Mayou RA, Peveler RC, Neil HA. Poor prognosis of young adults with type 1 diabetes: a longitudinal study. Diabetes Care. 2003 Apr;26(4):1052-7. doi: 10.2337/diacare.26.4.1052. PMID 12663572
- [Background] White NH, Cleary PA, Dahms W, Goldstein D, Malone J, Tamborlane WV; Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Interventions and Complications (EDIC) Research Group. Beneficial effects of intensive therapy of diabetes during adolescence: outcomes after the conclusion of the Diabetes Control and Complications Trial (DCCT). J Pediatr. 2001 Dec;139(6):804-12. doi: 10.1067/mpd.2001.118887. PMID 11743505
- [Background] Channon S, Smith VJ, Gregory JW. A pilot study of motivational interviewing in adolescents with diabetes. Arch Dis Child. 2003 Aug;88(8):680-3. doi: 10.1136/adc.88.8.680. PMID 12876161
- [Background] Rubak S, Sandbaek A, Lauritzen T, Christensen B. Motivational interviewing: a systematic review and meta-analysis. Br J Gen Pract. 2005 Apr;55(513):305-12. PMID 15826439
- [Background] Service FJ, Molnar GD, Rosevear JW, Ackerman E, Gatewood LC, Taylor WF. Mean amplitude of glycemic excursions, a measure of diabetic instability. Diabetes. 1970 Sep;19(9):644-55. doi: 10.2337/diab.19.9.644. No abstract available. PMID 5469118
- [Background] Valerio G, del Puente A, Esposito-del Puente A, Buono P, Mozzillo E, Franzese A. The lumbar bone mineral density is affected by long-term poor metabolic control in adolescents with type 1 diabetes mellitus. Horm Res. 2002;58(6):266-72. doi: 10.1159/000066441. PMID 12446989
- [Background] Sarkola T, Redington A, Keeley F, Bradley T, Jaeggi E. Transcutaneous very-high-resolution ultrasound to quantify arterial wall layers of muscular and elastic arteries: validation of a method. Atherosclerosis. 2010 Oct;212(2):516-23. doi: 10.1016/j.atherosclerosis.2010.06.043. Epub 2010 Jul 7. PMID 20673898
- [Derived] Pulkkinen MA, Tuomaala AK, Hero M, Gordin D, Sarkola T. Motivational Interview to improve vascular health in Adolescents with poorly controlled type 1 Diabetes (MIAD): a randomized controlled trial. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001216. doi: 10.1136/bmjdrc-2020-001216. PMID 32723754